CLINICAL TRIAL: NCT04408482
Title: Does Pancreatic Stent Decrease the Risk of Pancreatitis After Pancreatic Sphincterotomy for Difficult Cannulation?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Andrea Tenca, Principal investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3509/2019
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pancreatic sphincterotomy (Active Comparator): Pancreatic sphincterotomy performed in difficult cannulation
  Interventions: Device: Biliary cannulation
- Pancreatic sphincterotomy + pancreatic stent (Active Comparator): Pancreatic sphincterotomy performed in difficult cannulation + pancreatic stent placement
  Interventions: Device: Biliary cannulation

INTERVENTIONS:
Device: Biliary cannulation — Cannulation of biliary duct by sphincterotome

SUMMARY:
The purpose of the study is to compare the risk of PEP after pancreatic sphincterotomy performed for difficult cannulation in a group of patients with and in a group of patients without placement of a prophylactic pancreatic stent. The definition of difficult cannulation is defined according to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with naïve papilla presenting to ERCP with indication of common bile duct (CBD) cannulation will be considered to the study.

Exclusion Criteria:

* Exclusion criteria are age below 18 years, acute pancreatitis and no consent to the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis rate | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki Univeristy Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided